CLINICAL TRIAL: NCT00410332
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study for Evaluating the Efficacy of the Homeopathic Remedy Traumeel S on Pain Reduction Following Tonsillectomy in Adult Patients.
Brief Title: Traumeel for Post-Tonsillectomy Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32/6
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Post-Tonsillectomy
Keywords: tonsillectomy; pain; homeopathy; Traumeel
MeSH Terms: conditions — Pain | interventions — Traumeel S

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Active Comparator): TRAUMEEL S
  Interventions: Drug: Traumeel S
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traumeel S — homeopathic remedy
  Arms: A
Drug: Placebo — placebo drug, identical in size, form and taste as treatment remedy
  Arms: B

SUMMARY:
Tonsillectomy is one the most common procedures in ear, nose and throat (ENT) medicine. Following surgery patients suffer from severe pain and difficulty on swallowing, while analgesic treatment has limited efficacy and potential adverse effects such as increased bleeding with NSAIDs. Traumeel S is a homeopathic complex remedy used primarily in Europe for the treatment of pain and inflammation. It contains a number of plants and minerals at high dilutions (between 1x10-2 to 1x10-8), and has been shown to exhibit anti-inflammatory properties such as cytokine inhibition in human T cells, monocytes and gut epithelial cells. Clinical studies have found Traumeel S reduces post-chemotherapy stomatitis, as well as post-surgical inflammation and pain following orthopedic procedures.

The purpose of this study is to examine the effect of Traumeel S on post-tonsillectomy pain in adult patients. The study group will consist of 20 patients age 18 years of age and older following elective tonsillectomy. These patients will be randomly assigned to receive treatment with either true Traumeel S remedies or placebo. One ampule of Traumeel S (or placebo) will be sprayed over the resected area immediately following surgery. Two Traumeel S (or placebo) tablets will be taken subsequently 4 times daily (Total: 8 tablets per day)until no analgesics are required for 2 consecutive days, or until Day 14 (whichever comes first). Patients will be allowed to take dipyrone (Optalgin) 500mg tablets on an as-needed basis, for up to 14 days postoperatively. At the end of this period, a thorough ENT examination will be done.

The primary parameter to be evaluated in the study will be postoperative pain, as registered on a numerical pain rating scale (NRS), to be filled prior to surgery. In the post-anesthesia care unit (PACA) the NRS will be filled out again, this time for pain at rest and then again for pain upon swallowing - at 1, 2, 3,4 and 24 hours postoperatively. Secondary parameters to be evaluated are: analgesic use (dipyrone); post-operative bleeding (quantified on a scale of 1-4); nocturnal awakenings; time to resumption of eating and return to normal activity; cytokine levels (CRP, IL-6) at 36 hours postoperative; and side effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Recurrent tonsillitis or obstructive tonsillar hypertrophy requiring tonsillectomy.

Exclusion Criteria:

* Elective or emergency tonsillectomy for a reason other than those listed above.
* History of peritonsillar abscess, or need for additional ENT procedures (adenoidectomy, uvulectomy)
* Pregnancy, breastfeeding
* Asthma, Epilepsy
* Concurrent illness with impairment of wound-healing (diabetes, vascular disease)
* allergy or contraindication to use of protocol medication (dipyrone)
* inability to comply with the protocol conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain, as registered on the NRS | 14d

SECONDARY OUTCOMES:
analgesic use (dipyrone) | 14d
post-operative bleeding (quantified on a scale of 1-4) | 14d
nocturnal awakenings | 14d
time to resumption of eating and return to normal activity | 14d
cytokine levels (CRP, IL-6) at 36 hours postoperative | 14d
side effects of the treatment. | 14d

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Dept. of Ear, Nose and Throat Medicine, Shaare Zedek Medical Center, Jerusalem, Israel